CLINICAL TRIAL: NCT00097214
Title: A Phase II Trial of Carboplatin Plus Cetuximab for the Treatment of Stage IIIb/IV Non-Small Cell Lung Cancer
Brief Title: Carboplatin Plus Cetuximab for Treatment of Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-081
Record Dates: First submitted 2004-11-18; First posted 2004-11-19 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Non-small; Lung; IIIB; IV; Carboplatin; Cetuximab; Stage IIIB non-small cell lung cancer; Stage IV non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cetuximab 400 mg/m2 IV on Day 1, followed by weekly doses of 250 mg/m2 IV beginning on Day 8. Carboplatin AUC= 6 IV will be given on the first day of each 3-week cycle, beginning on Day 8.
  Therapy will continue for four cycles (12 weeks)for combination therapy
  Interventions: Drug: Carboplatin; Biological: Cetuximab

INTERVENTIONS:
Drug: Carboplatin — AUC= 6 IV will be given on the first day of each 3-week cycle, beginning on Day 8.
  Other Names: Paraplatin
Biological: Cetuximab — 400 mg/m2 IV on Day 1, followed by weekly doses of 250 mg/m2 IV beginning on Day 8.
  Other Names: erbitux

SUMMARY:
This is a phase II study in previously untreated subjects with histologically or cytologically proven stage IIIB/IV NSCLC designed to determine the efficacy of first line treatment with carboplatin and cetuximab.

DETAILED DESCRIPTION:
Lung cancer is the second most common cancer diagnosed for both genders in the United States. Approximately 173,770 new cases are estimated for 2004. It is the leading cause of cancer deaths in both men and women, with approximately 160,440 deaths estimated for 2004. Prognosis for many is poor if not diagnosed at an early stage, and therapy for advanced disease is limited. The study will test carboplatin in combination with a newly approved drug called cetuximab, which is continuing to be tested in colorectal cancer and other cancers. Cetuximab is a monoclonal antibody, which is believed to work by attaching to an epidermal growth factor receptor (EGFR) on tumor cells and thereby blocking tumor cells from reproducing. It is an antibody to the EGFR. Fifty percent of lung cancers overexpress EGFR.

Rationale:

The present study is built upon the data from the described studies, incorporating cetuximab into a regimen of single-agent carboplatin. Previous data suggest that single agent carboplatin is active in NSCLC. The addition of biologic therapy with the anti-EGFR agent cetuximab to carboplatin will presumably maximize the therapeutic index while keeping toxicity to a minimum in patients with Stage IIIB/IV NSCLC.

Research Hypothesis:

The population being studied in this trial is subjects with previously untreated Stage IIIB or IV NSCLC. The research hypothesis is that these subjects will achieve a response (based on RECIST criteria) to therapy with the combination of carboplatin and cetuximab.

ELIGIBILITY:
INCLUSION CRITERIA:

To be eligible for the study, subjects must fulfill all of the following criteria.

* Subjects must have signed an approved informed consent.
* Subjects with histologically or cytologically documented stage IIIB (supraclavicular lymph node, high neck node, or pleural effusion involvement) or IV NSCLC. Disease must be newly diagnosed or recurrent at least 1 year post adjuvant therapy.
* Subjects with measurable disease.
* Subjects with ECOG performance status 0-1.
* If diagnostic tissue or slides are available for a subject, these must be submitted for testing of EGFR status.
* Subjects with asymptomatic brain metastasis are eligible; however, they must have completed radiotherapy/radiosurgery at least 2 weeks prior to enrollment. Radiotherapy must have been completed >2 weeks prior to enrollment and the subject must have recovered from all adverse effects of prior radiotherapy. No previous irradiation to the only area of measurable disease. New lesions that developed in a previously irradiated area will be allowed.
* Subjects ≥18 years of age.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea ≥12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level >35mIU/mL]. Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication.

Physical and Laboratory Test Findings

* Subjects with adequate hematologic function defined as: ANC ≥1,500/mm 3 ; WBC

  ≥3,000/mm 3 ; platelets ≥100,000/mm 3 ; and hemoglobin ≥9 g/dL.
* Subjects with adequate hepatic function defined as: total bilirubin ≤1.5 x upper limit of normal (ULN) or AST ≤2.5 x ULN.
* Subjects with adequate renal function defined as a serum creatinine level ≤1.5 mg/dL or a creatinine clearance ≥60 cc/minute.

EXCLUSION CRITERIA:

Any of the following criteria will make the subject ineligible to participate in this study:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study. Subjects who are men must also agree to use effective contraception.
* WOCBP using a prohibited contraceptive method.
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Subjects who have had prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the subject has been disease-free for 5 years.
* Subjects with significant history of cardiac disease, i.e., uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure, cardiomyopathy with decreased ejection fraction, myocardial infarction within the past year, or cardiac ventricular arrythmias requiring medication.
* Subjects with an uncontrolled seizure disorder, or active neurological disease.
* Subjects with symptomatic brain metastasis.

Prohibited Therapies and/or Medications

* Subjects who have received prior systemic chemotherapy. Subjects with no more than one prior adjuvant regimen for initially diagnosed disease are eligible for the study.
* Subjects with a history of prior cetuximab or other therapy that specifically and directly targets the EGFR pathway.
* Subject with prior severe reaction to a monoclonal antibody.
* Subjects with prior erythropoietin (i.e., Epogen, Procrit) treatment
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall response rate | Every six months

SECONDARY OUTCOMES:
To evaluate the proportion of subjects with progression free survival (median and 6 months) | Every six months
To evaluate survival times (median and 1-year) | Every six months
To evaluate the toxicity profiles of the treatment regimen | Every 12 weeks
To evaluate symptom response rate using the Lung Cancer Subscale (LCS) of the FACT-L | Every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (8):
- United States (8):
  - ImClone Investigational Site, Bentonville, Arkansas
  - ImClone Investigational Site, Tucker, Georgia
  - ImClone Investigational Site, Evanston, Illinois
  - ImClone Investigational Site, Louisville, Kentucky
  - ImClone Investigational Site, Chapel Hill, North Carolina
  - ImClone Investigational Site, Fayetteville, North Carolina
  - ImClone Investigational Site, Langhorne, Pennsylvania
  - ImClone Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Bradford DS, Socinski MA, LaRocca RV, Hensing TA, Bordoni RE. Phase II trial of carboplatin plus cetuximab for the treatment of Stage IIIB/IV non-small cell lung cancer (NSCLC). J Clin Oncol, 2007 ASCO Annual Meeting Proceedings Part I. Vol 25, No. 18S (June 20 Supplement), 2007: 18005.